CLINICAL TRIAL: NCT06219603
Title: Knowledge and Awareness About Inflammatory Articular Diseases: A Cross Sectional Survey From a Syrian Population
Brief Title: Knowledge and Awareness About Inflammatory Articular Diseases
Status: Completed | Type: Observational
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Diaa Haj Ali, medical doctor Diaa Haj Ali, Syrian Private University
Other Study IDs: IRB; CW 855.1-12-2021
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Articular Diseases
Keywords: knowledge; Awareness; Inflammatory Articular Diseases; Syrian population
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- excellent: participants who answered on > 80 % of the questioned correctly
  Interventions: Other: survey
- good: participants who answered on 61 - 80 % of the questioned correctly
  Interventions: Other: survey
- average: participants who answered on 41 - 60 % of the questioned correctly
  Interventions: Other: survey
- bad: participants who answered on 21 - 40 % of the questioned correctly
  Interventions: Other: survey
- very bad: participants who answered on <=20 % of the questioned correctly
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — questions around socio-demographic information, including age, sex, marital status, residency, education level, and employment status. After that, specific questions were asked to measure the level of knowledge and awareness about rheumatic diseases

SUMMARY:
The manuscript describes the level of knowledge and awareness about Inflammatory Articular Diseases in a Syrian population. we found that awareness of Inflammatory Articular Diseases is mostly bad and very bad in our sample. Also, we showed how the level of awareness changes due to the change of many factors such as (sex, age, residency, education, marital status, and others ).

Our community-based survey was the first conducted in Syria. we have included a total of 641 participants who were directed to the first part of the survey to complete questions around socio-demographic data and awareness questions about Inflammatory Articular Diseases. We ranked our participants into five levels: excellent, good, average, bad, and very bad.

Finally, we compared our results with other 4 original published studies, and we found many Boolean points of similarity and many other inspiring points of difference.

ELIGIBILITY:
Inclusion Criteria:

* all participants older than 18 years and younger than 70

Exclusion Criteria:

* Non-Syrians

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A random sample from all segments of the Syrian population
Sampling Method: Non-Probability Sample
Enrollment: 641 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
knowledge about Inflammatory Articular Diseases | 1 year
  We ranked level of knowledge and awareness about Inflammatory Articular Diseases into five levels: excellent, good, average, bad, and very bad.
  higher knowledge level scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, syrian private University, Syria, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided